CLINICAL TRIAL: NCT00796354
Title: A Phase IIIb/IV, Multi-centre, Double-blind, Randomised, Placebo-controlled Parallel Group Study to Compare the Efficacy and Safety of Movicol® With Placebo in Patients With Constipation Associated With Irritable Bowel Syndrome (IBS)
Brief Title: Constipation Associated With Irritable Bowel Syndrome (IBS-C)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Dr Mike Geraint, Norgine Pharmaceuticals Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NRL920-01/2008 (IBSc)
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Constipation
Keywords: Constipation; Irritable Bowel Syndrome
MeSH Terms: conditions — Constipation; Irritable Bowel Syndrome | interventions — Polyethylene Glycols; Sodium Chloride; Sodium Bicarbonate; Potassium Chloride; acetosulfame; Sugars; Sucrose; lime

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NRL920 (Active Comparator)
  Interventions: Drug: MOVICOL
- Placebo (Placebo Comparator)
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: MOVICOL — sealed laminated sachet, 1 - 3 sachets daily for 4 weeks
  Other Names: Macrogol (PEG) 3350; sodium chloride; sodium bicarbonate; potassium chloride; acesulfame potassium; lemon-lime flavouring
  Arms: NRL920
Drug: Sugar Pill — sealed laminated sachet, 1 - 3 sachets daily for 4 weeks
  Other Names: Sucrose; lemon and lime flavour
  Arms: Placebo

SUMMARY:
Multi-centre, double-blind, randomised, placebo-controlled, parallel group study.

DETAILED DESCRIPTION:
Patients will be treated for 28 days, with clinical assessments carried out over 2 visits. Follow-up will be performed via telephone at a specific interval during the study to determine the outcome of unresolved AEs, any new drug-related AEs or any pregnancies. During the run-in period and the treatment phase, patients are prohibited from taking prescription or over the counter (OTC) laxative medication or constipating medications. Prescription and OTC medications not related to constipation are permitted and must be fully documented, but any changes (e.g., dosage, regimen) are to be limited as much as possible.

ELIGIBILITY:
Inclusion Criteria:

* Male and females aged 18 to 80 years inclusive.
* Written informed consent obtained.
* Females of child-bearing potential must employ an adequate method of contraception and must undergo a pregnancy test at Randomisation Visit.
* Willing, able and competent to complete the entire study and comply with study instructions.
* Patients > 50 years old have to have undergone a colonoscopy or computerised tomography (CT) after the onset of their IBS-C symptoms or within the last 5 years.
* Patient has diagnosed IBS-C using Rome III criteria for the last 3 months, with symptom onset at least 6 months prior to diagnosis.

Exclusion Criteria:

* History or evidence of organic disease in the large bowel, intestinal perforation or obstruction due to structural or functional disorder of the gut wall, ileus, severe inflammatory conditions of the intestinal tract such as Crohn's disease, complicated diverticulitis, ulcerative colitis, toxic megacolon and occlusive or subocclusive syndrome.
* Abdominal pain of unknown cause, not related to IBS.
* Previous major abdominal surgery.
* IBS subtype other than IBS-C.
* Known allergy to polyethylene glycol (PEG) 3350 or known hypersensitivity to any of the active substances.
* Laxative, drug or alcohol abuse (recent history or within previous 12 months).
* Pregnant or lactating females.
* Severe or acute disease within 2 weeks prior to the start of the study.
* Patients with type I or II diabetes.
* Use of other investigational drugs, prescribed or OTC medications affecting gastrointestinal function such as anticholinergics, prokinetics, drugs affecting motility, anthraquinones, opioids,ondansetron or other 5-HT3 antagonists.
* Incomplete Patient Diary Card during the run-in period.
* The occurrence of diarrhoea* during the run-in period.
* Patients with abnormal laboratory tests, proctoscopy /abdominal ultrasound, colonoscopy, sigmoidoscopy or CT that requires further investigation.
* Patients with any condition, which, in the Investigator's may put the patient at significant risk, may confound the study results, or may interfere significantly with the results of the study.
* Participation in another clinical study of drugs or devices parallel to or less than 1 month before study entry, or previous participation in this study.
* Employees of the Investigator or study site with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, as well as family members of the employees or the Investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2008-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy and safety of Movicol® versus placebo in the relief of constipation associated with IBS. | April 2009

SECONDARY OUTCOMES:
To evaluate the effect of treatment on other symptoms of IBS. | April 2009
To evaluate the effect of treatment on patient's Quality Of Life (QOL). | April 2009

CONTACTS AND LOCATIONS:
Overall Officials: Roger Chapman, MD, Principal Investigator — Oxford University Hospitals NHS Trust; Mike Geraint, MD, Study Director — Norgine Pharmaceuticals Ltd
Locations (21):
- Czechia (3):
  - Gastroenterologie s.r.o., Hradec Králové
  - EGK.s.r.o, Sanatorium sv. Anny, Prague
  - Orlickoustecká Nemocnice a.s., Ústi Nad Orlicí
- France (3):
  - Hôpital Hotel Dieu, Clermont-Ferrand
  - Hôpital Archet II, Nice
  - Hôpital Charles Nicolles, Rouen
- Germany (3):
  - Martin-Luther-Krankenhaus-Betriebs-GmbH, Berlin
  - Gastroenterologische Gemeinschaftspraxis, Münster
  - Facharztpraxis für Innere Medizin, Wiesbaden
- Italy (4):
  - Policlinico S. Orsola Malpighi, Bologna
  - Università degli Studi di Genova, Genova
  - Università degli Studi di Palermo, Palermo
  - Università La Sapienza, Roma
- Poland (4):
  - Slaskie Centrum Osteoporozy, Katowice
  - Prosen SMO, Warsaw
  - Centrum Onkologii ul.Rentgena 5, Warsaw
  - Katedra i Klinika Gastroenterologii i Hepatologii, Wroclaw
- Sweden (2):
  - Sodra Alvsborgs Hospital (SAS), Borås
  - Karolinska University Hospital Solna, Stockholm
- United Kingdom (2):
  - St Marks Hospital, Harrow
  - John Radcliffe Hospital, Oxford

REFERENCES:
- [Background] Attar A, Lemann M, Ferguson A, Halphen M, Boutron MC, Flourie B, Alix E, Salmeron M, Guillemot F, Chaussade S, Menard AM, Moreau J, Naudin G, Barthet M. Comparison of a low dose polyethylene glycol electrolyte solution with lactulose for treatment of chronic constipation. Gut. 1999 Feb;44(2):226-30. doi: 10.1136/gut.44.2.226. PMID 9895382